CLINICAL TRIAL: NCT06157892
Title: A Phase 1b/2 Open-Label Study of Disitamab Vedotin in Combination With Other Anticancer Therapies in Solid Tumors
Brief Title: A Study of Disitamab Vedotin With Other Anticancer Drugs in Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNDV-004; C5731004 (Other: Alias Study Number); 2023-507555-29-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms; Gastroesophageal Junction Adenocarcinoma; HER2 Low Breast Neoplasms; HER2 Positive Breast Neoplasms; Stomach Neoplasms; Triple Negative Breast Neoplasms; Metastatic Breast Cancer; Metastatic Gastric Cancer; Advanced Breast Cancer; Advanced Gastric Cancer
Keywords: Breast Cancer; Gastric Cancer; GC; GEJ; HER2-Low Breast Cancer; HER2-Positive Breast Cancer; Seattle Genetics
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Triple Negative Breast Neoplasms | interventions — disitamab vedotin; RC48 antibody; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation - Previously treated advanced GC/GEJC or breast cancer (Experimental): disitamab vedotin + tucatinib
  Interventions: Drug: disitamab vedotin; Drug: tucatinib
- Dose Optimization - HER2-low and HER2+ LA/mBC (Experimental): disitamab vedotin + tucatinib
  Interventions: Drug: disitamab vedotin; Drug: tucatinib
- Dose Optimization - HER2-low and HER2+ LA/mGC/GEJC (Experimental): disitamab vedotin + tucatinib
  Interventions: Drug: disitamab vedotin; Drug: tucatinib
- Dose Expansion - HER2-low LA/mBC (Experimental): disitamab vedotin + tucatinib
  Interventions: Drug: disitamab vedotin; Drug: tucatinib
- Dose Expansion - HER2+ LA/mBC (Experimental): disitamab vedotin + tucatinib
  Interventions: Drug: disitamab vedotin; Drug: tucatinib
- Dose Expansion - HER2-low LA/mGC/GEJC (Experimental): disitamab vedotin + tucatinib
  Interventions: Drug: disitamab vedotin; Drug: tucatinib
- Dose Expansion - HER2+ LA/mGC/GEJC (Experimental): disitamab vedotin + tucatinib
  Interventions: Drug: disitamab vedotin; Drug: tucatinib

INTERVENTIONS:
Drug: disitamab vedotin — Given into the vein (IV; intravenous)
  Other Names: RC48, RC48-ADC
Drug: tucatinib — 300mg given twice daily by mouth (orally)
  Other Names: TUKYSA, ONT-380, ARRY-380

SUMMARY:
This clinical trial is studying solid tumor cancers. A solid tumor is one that starts in part of your body like your lungs or liver instead of your blood. Once they've grown bigger in one spot or spread to other parts of the body, they're harder to treat. This is called advanced or metastatic cancer.

Participants in this study must have breast cancer or gastric cancer. Participants must have tumors that have HER2 on them. This allows the cancer to grow more quickly or spread faster. There are few treatment options for patients with advanced or metastatic solid tumors that express HER2.

This clinical trial uses an experimental drug called disitamab vedotin (DV). Disitamab vedotin is a type of antibody drug conjugate or ADC. ADCs are designed to stick to cancer cells and kill them.

This clinical trial uses a drug called tucatinib, which has been approved to treat cancer in the United States and some other countries. This drug is sold under the brand name TUKYSA®.

This study will test how safe and how well DV with tucatinib works for participants with solid tumors. This study will also test what side effects happen when participants take these drugs. A side effect is anything a drug does to the body besides treating the disease.

DETAILED DESCRIPTION:
This clinical trial is to evaluate disitamab vedotin in combination with tucatinib in subjects with LA/metastatic breast cancer or gastric cancer/GEJC that express HER2. The study has a dose escalation phase evaluating disitamab vedotin plus tucatinib followed by a dose optimization phase. The 2 dose levels identified in the dose escalation phase will be assessed in the optimization phase for both safety and efficacy in HER2-expressing LA/mBC and LA/mGC/GEJC. Once the safety and efficacy profile of disitamab vedotin plus tucatinib has been established and a disitamab vedotin dose with the optimum benefit/risk ratio has been determined the disitamab vedotin plus tucatinib combination therapy will be evaluated in an expansion phase with 4 expansion cohorts in subjects with HER2-low LA/mGC/GEJC, HER2+ LA/mGC/GEJC, HER2-low LA/mBC, and HER2+ LA/mBC.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Measurable disease according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1

Dose Escalation and Optimization Phase Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma or breast carcinoma
* Locally-advanced, unresectable, or metastatic stage
* Must have experienced disease progression on or after standard of care therapies or be intolerant of standard of care therapies.

Cohort A (HER2-Low Breast Cancer) Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of breast carcinoma
* Locally-advanced, unresectable, or metastatic stage
* HER2-low status determined by most recent local assessment (IHC 1+ or IHC 2+/ISH-negative)
* Prior therapies requirements

  * No more than 3 prior systemic cytotoxic chemotherapy regimens (including ADCs) for LA/mBC.
  * Participants with known BRCA mutation must have received a PARP-inhibitor where available and not medically contraindicated
  * Have progression on or after, or intolerant to, T-DXd, sacituzumab govitecan, or other topoisomerase I inhibitor therapies, if available as local standard of care therapy
  * Participants with HR+ tumors must have intolerance to endocrine therapy or endocrine therapy refractory disease:

    * Progressed on ≥2 lines of endocrine therapy for LA/mBC AND had received a CDK4/6 inhibitor in the adjuvant or metastatic setting OR
    * Progressed on 1 line of endocrine therapy for LA/mBC AND had a relapse while on adjuvant endocrine therapy after definitive surgery for primary tumor AND had received a CDK4/6 inhibitor in the adjuvant or advanced setting
  * Participants with HR negative, HER2-low and PD-L1-positive (CPS 10 or greater) tumors must have received pembrolizumab with chemotherapy if available as local standard of care therapy.
  * Participants with HR negative, HER2-low and PD-L1-positive (CPS 10 or greater) tumors must have received pembrolizumab (or other PD-(L)1 inhibitor) with chemotherapy if available as local standard of care therapy and not medically contraindicated.

Cohort B (HER2+ Breast Cancer) Inclusion Criteria

* Histologically or cytologically confirmed diagnosis breast carcinoma
* Locally-advanced, unresectable, or metastatic stage
* HER2+ status determined by most recent local assessment (IHC 3+ or IHC 2+/ISH+)
* Participants must have:

  * Received prior trastuzumab, pertuzumab and a taxane if available as local standard of care therapy for advanced disease.
  * Have progression on or after, or intolerant to, T-DXd or other topoisomerase I inhibitor therapies
  * No more than 3 prior systemic cytotoxic chemotherapy regimens (including ADCs) for LA/mBC

Cohort C (HER2-Low Gastric or Gastroesophageal Junction Adenocarcinoma) Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma
* Locally-advanced, unresectable, or metastatic stage
* HER2-low expression defined as IHC 1+ or IHC 2+/ISH-negative determined by most recent local assessment
* Willing and able to provide archival or newly obtained formalin-fixed paraffin-embedded (FFPE) tumor tissue blocks
* Participants must have received:

  * Prior systemic therapy with platinum, fluorouracil, or taxane for locally advanced unresectable or metastatic disease
  * Progression within 6 months of last dose of (neo)adjuvant cytotoxic chemotherapy is considered as 1 line of systemic therapy for LA/mGC/GEJC
  * Prior anti-PD-(L)1 therapy is allowed
  * No more than 2 prior systemic cytotoxic chemotherapy regimens (including ADC) for LA/mGC/GEJC
* Must not have received prior treatment with HER2 directed therapy

Cohort D (HER2+ LA/mGC/GEJC) Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma
* Locally-advanced, unresectable, or metastatic stage
* HER2+ status determined by most recent local assessment (IHC 3+ or IHC 2+/ISH+)
* Participants must have:

  * Received prior trastuzumab plus fluoropyrimidine and platinum containing chemotherapy if no contraindication.
  * Prior T-DXd treatment is allowed
  * Prior PD1 inhibitor therapy is allowed
  * No more than 2 prior systemic cytotoxic chemotherapy regimens (including ADCs) for LA/mGC/GEJC

Exclusion Criteria:

* Known hypersensitivity to any excipient contained in the drug formulation of disitamab vedotin or tucatinib
* Prior therapy with ADCs with MMAE payload
* Prior therapy with tucatinib
* Active CNS and/or leptomeningeal metastasis.
* Participants who have received prior systemic anticancer treatment including investigational agents within 4 weeks prior to first dose of study treatment
* History of other invasive malignancy within 3 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy.
* Unable to swallow oral tablets or capsules or any significant GI disease which would preclude the adequate oral absorption of medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2029-07-28 (Estimated); Study Completion 2029-07-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) in dose escalation phase | Up to 28 days
Number of participants with adverse events (AEs) | Through 30 days after the last study treatment; approximately 5 years
  Any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of participants with laboratory abnormalities | Through 30-37 days after the last study treatment: approximately 5 years
Number of participants with dose alterations | Through 30-37 days after the last study treatment: approximately 5 years
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) by investigator assessment | Approximately 3 years
  The proportion of participants with confirmed response (CR) or partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Duration of response (DOR) per RECIST v1.1 by investigator assessment | Approximately 5 years
  The time from start of the first documentation of objective tumor response of CR or PR (that is subsequently confirmed) to the first documentation of progressive disease (PD) per RECIST v1.1, or to death due to any cause
Disease control rate (DCR) per RECIST v1.1 by investigator assessment | Approximately 5 years
  The proportion of participants with stable disease (SD) or confirmed CR or PR according to RECIST v1.1.
Progression free survival (PFS) per RECIST v1.1 by investigator assessment | Approximately 5 years
  The time from the start of any study treatment (or randomization date for participants in dose optimization phase) to the first documentation of disease progression per RECIST v1.1 or death due to any cause.
Overall survival (OS) | Approximately 5 years
  The time from the start of any study treatment (or randomization date for participants in dose optimization phase) to the date of death due to any cause.
Pharmacokinetic (PK) parameter - Maximum concentration (Cmax) | Through 30-37 days after the last study treatment; approximately 5 years
PK parameter - Area under the concentration-time curve to the time of the last quantifiable concentration (AUClast) | Approximately 1 month
Incidence of anti-drug antibodies (ADAs) against disitamab vedotin | Through 30-37 days after the last study treatment; approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (134):
- United States (79):
  - Banner-University Medical Center Tucson Campus, Tucson, Arizona
  - The University of Arizona Cancer Center-North Campus Pharmacy, Attn: Kelly Myrdal, Tucson, Arizona
  - University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - The University of Arizona Cancer Center-Main, Tucson, Arizona
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - UC Irvine Medical Center, Orange, California
  - University of California, San Francisco | HDFCCC - Hematopoietic Malignancies, San Francisco, California
  - UCLA Department of Medicine - Hematology & Oncology, Santa Monica, California
  - UCLA Hematology/Oncology - Parkside, Santa Monica, California
  - Colorado West Healthcare System, dba Community Hospital, Grand Junction, Colorado
  - Colorado West Healthcare, dba Grand Valley Oncology, Grand Junction, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - The Whittingham Cancer Center / Norwalk Hospital, Norwalk, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center - International Plaza, Tampa, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt McKinley Hospital, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Georgia Cancer Specialists - Athens, Athens, Georgia
  - Georgia Cancer Specialists - Annex, Atlanta, Georgia
  - Atlanta Cancer Care - Atlanta, Atlanta, Georgia
  - Georgia Cancer Specialists-Northside, Atlanta, Georgia
  - Northside Hospital, Inc.- Central Research Department, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Georgia Cancer Specialists - Blairsville, Blairsville, Georgia
  - Georgia Cancer Specialists - Canton, Canton, Georgia
  - Atlanta Cancer Care - Cumming, Cumming, Georgia
  - Georgia Cancer Specialists - Cumming, Cumming, Georgia
  - Georgia Cancer Specialists - Decatur, Decatur, Georgia
  - Suburban Hematology-Oncology Associates - Duluth, Duluth, Georgia
  - Suburban Hematology-Oncology Associates- Lawrenceville, Lawrenceville, Georgia
  - Georgia Cancer Specialists - Macon, Macon, Georgia
  - Georgia Cancer Specialists - Marietta, Marietta, Georgia
  - Memorial Hospital, Shiloh, Illinois
  - Siteman Cancer Center - Shiloh, Shiloh, Illinois
  - Massachusetts General Hospital., Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute- Chestnut Hill, Newton, Massachusetts
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Saint Luke's Cancer Institute LLC, Kansas City, Missouri
  - Saint Luke's Hospital Investigational Pharmacy, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth., Middletown, New Jersey
  - MSK Bergen., Montvale, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - MSK Commack., Commack, New York
  - MSK Westchester., Harrison, New York
  - Investigational Drug Service, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - Main Hospital, New York, New York
  - MSK Nassau., Uniondale, New York
  - Zangmeister Cancer Center, Columbus, Ohio
  - Saint Francis Hospital / Bon Secours - South Carolina, Greenville, South Carolina
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute, Nashville, Tennessee
  - Parkland Health and Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center-Simmons Cancer Center Pharmacy, Dallas, Texas
  - University of Texas Southwestern Medical Center Simmons Cancer Center - Redbird, Dallas, Texas
  - University of Texas Southwestern Medical Center Clinical Lab-Zale Lipshy University Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center-William P. Clements Jr. University Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Southwestern Simmons Cancer Center - Fort Worth, Fort Worth, Texas
  - University of Texas Southwestern Medical Center Simmons Cancer Center - Richardson/Plano, Richardson, Texas
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center / Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin
- Australia (6):
  - Peninsula & South Eastern Hematology and Oncology Group (PASO), Frankston, Victoria
  - Slade Pharmacy Frankston, Frankston, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Slade Health, Mount Waverley, Victoria
  - Peninsula & South Eastern Hematology and Oncology Group (PASO), Frankston
  - Peter MacCallum Cancer Centre, Melbourne
- Canada (4):
  - BC Cancer Kelowna., Kelowna, British Columbia
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
- Germany (4):
  - Charité Universitätsmedizin Berlin, Campus Benjamin Franklin (CBF), Berlin
  - Universitatsklinikum Essen, Essen
  - Heidelberg University Hospital and German Cancer Research Center, Heidelberg
  - Klinikums rechts der Isar der TU München, München
- Italy (8):
  - A.O.U. Federico II, Napoli, Campania
  - Azienda Ospedaliera Universitaria (AOU) Federico II, Napoli, Campania
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale., Napoli, Campania
  - Istituto Europeo di Oncologia, Milan, Lombardy
  - Niguarda Ca' Granda Hospital, Milan, Lombardy
  - Humanitas Istituto Clinico Catanese, Misterbianco (CT), Sicily
  - Azienda Ospedaliera Universitaria Integrata di Verona., Verona, Veneto
  - A.O.U. Federico II- U.O.C. Diagnostica per lmmagini e Radioterapia, Napoli
- South Korea (10):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Dong-A University Hospital, Busan, Other
  - National Cancer Center, Goyang-si, Other
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon
- Spain (10):
  - Quirén Salud Barcelona, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - CETIR Grup Medic, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Grupo Hospitalario QuironSalud, Erandio Bizkaia
  - Farmacia-Ensayos. Planta S - Hospital Universitario HM Sanchinarro-CIOCC-START Madrid, Madrid
  - START Madrid-CIOCC_Hospital HM Sanchinarro, Madrid
  - Ecg Medica Sl, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (5):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (8):
  - The Royal Marsden Hospital, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - St Bartholomew's Hospital, London
  - The Royal Marsden Hospital, London
  - The Royal Marsden NHS Foundation Trust (RM), London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNDV-004